CLINICAL TRIAL: NCT04939038
Title: Timing of Revascularization in Patients With Diabetic Foot Ulcer and Non-critical Peripheral Artery Disease: a Randomized, Controlled Trial
Brief Title: Timing of Revascularization in Patients With Diabetic Foot Ulcer and Non-critical Peripheral Artery Disease
Acronym: DIFU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High pre-screening failure and insufficient recruited patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1495 DIFU
Record Dates: First submitted 2021-06-23; First posted 2021-06-25 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Revascularization; Lower extremity arterial disease; Non-critical peripheral artery disease
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Standard wound care for diabetic wound ulcer
  Interventions: Procedure: Standard wound care
- Immediate revascularization (Experimental): Patient will have revascularization 0 - 7 days after initial wound assessment and then receive standard wound care for diabetic wound ulcer
  Interventions: Procedure: Revascularization; Procedure: Standard wound care

INTERVENTIONS:
Procedure: Revascularization — Depending on the condition of the patients, patients will have either endovascular or surgical revascularization
  Arms: Immediate revascularization
Procedure: Standard wound care — Standard wound care according to guidelines

SUMMARY:
This study investigates whether, compared to standard treatment, immediate restoration of blood flow (revascularization) can reduce complications and improve diabetic foot ulcer healing.

DETAILED DESCRIPTION:
Background: In approximately 80% of diabetes-related lower extremity amputations, patients suffer from a foot ulcer, often caused by lower extremity arterial disease. Due to lower extremity arterial disease (LEAD), diabetic patients with foot ulcers often require lower limb amputation. Achieving arterial supply (revascularization) to the ulcer is the most important factor in healing the diabetic foot ulcer and reduces the risk of amputation. The current standard of care recommends revascularization after six weeks in patients with low-grade arterial disease of the lower extremities and nonhealing foot ulcer. The aim of this study is to demonstrate that in patients with low grade arterial disease of the lower extremities and diabetic foot ulcers, immediate revascularization results in fewer cardiovascular problems and amputations, as well as improved ulcer healing, compared to the current standard of care.

Study procedure: After inclusion in the study, participants will be randomized into the control arm or the active arm. In the control arm standard wound care will be performed. In the active arm, revascularization will be performed on top of standard wound care within 7 days after randomization. Post-revascularization analysis on ankle- and toe pressure, laboratory analysis, and wound care team assessment and therapy will be performed 24 h post operation.

Follow up will be on 45, 90, 180 and 365 day for patients of both arms, where ankle- and toe pressure, laboratory analysis, and wound care team assessment and therapy will be performed.

Number of Participants: 240 participants in total, 120 per treatment arm

Study duration: 4 years

Study Centre(s): International multi-centre study with approximately 8-12 centres

Participating countries: Switzerland, Germany

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Patients that are at least 18 years old
* Patients that have at least one DFU(s) of ≥ 0.2 cm2 and ≤ 10 cm2 as assessed by the ruler method multiplying the greatest length and width of the ulcer after debridement to determine the surface area. The largest eligible ulcer (≤ 10 cm2) will be defined as index ulcer and the corresponding extremity as index limb (in case of multiple equally sized ulcers the following rules will apply: If on different feet, the dominant side and if on the same foot, the more peripheral one will be the index ulcer)
* Patients that have non-critical LEAD of the index leg, defined by a single non-invasive examination at screening:

  * Ankle brachial index (ABI) ≥ 0.5 and ≤ 0.9 AND absolute ankle pressure ≥ 50 mmHg OR
  * ABI > 0.9 OR incompressible ankle pressures AND toe brachial index (TBI) ≤ 0.7 AND absolute toe pressure ≥ 30 mmHg
* Patients on medical treatment for glycemic control with diagnosis of diabetes mellitus that was assessed by criteria as recommended by the guideline 2019 "ESC Guidelines on diabetes, pre-diabetes, and cardiovascular diseases developed in collaboration with the EASD". Or patient without medical treatment but diagnosed with diabetes mellitus via HbA1c.
* Patients with life expectancy > 12 months and without any disabilities due to end-stage cancer, heart failure, severe chronic obstructive pulmonary disease (COPD), or dementia

Exclusion Criteria:

* Critical limb ischemia of the index leg defined as ABI ≤ 0.4 (or absolute ankle pressure < 50 mmHg)
* No option to assess for toe pressure due to any reason at baseline if ABI > 0.9 or incompressible ankle pressures and patient inclusion is based on the toe pressure criteria.
* Need for major amputation
* Severe infection at the index foot according to IDSA classification
* Patient refuses minor amputation despite strong recommendation due to severe infection, necrosis or osteomyelitis at screening assessment
* Any revascularization procedure at the index leg within 3 months before randomization
* Positive urine or blood pregnancy test result, breast feeding or intention to become pregnant
* Non-compliance for any reason to procedures or study assessments (e.g. due to cognitive impairment or geographic distance)
* Participation in another drug study within the 30 days preceding or during the present study
* Untreated known antiphospholipid antibody syndrome and polycythaemia vera
* Known significant bleeding risk, or known coagulation disorder (INR > 3.0 and platelet count < 30,000/mm3) without any option to correct within 7 calendar days after initial wound assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with cardiovascular death | up to 12 months
Number of patients with non-fatal myocardial infarction or all-cause stroke | up to 12 months after randomization
Number of patients with major amputation | up to 12 months after randomization
Number of patients with Minor amputation | up to 12 months after randomization
Number of patients with missed diabetic foot ulcer healing | 90 days after randomization
  i.e. Incomplete epithelization of the index ulcer at 90 days
Number of patients with delayed diabetic foot ulcer healing | 45 days after randomization
  Reduction of wound size of less than 50% at 45 days

SECONDARY OUTCOMES:
Number of patients with new ulcer of the index foot | up to 12 months after randomization
Number of patients with all clinically-driven revascularizations at the index limb | up to 12 months after randomization
  excluding primary revascularization in the immediate re-vascularization group
Each component of the primary outcome individually | up to 12 months after randomization
  Primary outcome 1 to 6
Number of in-hospital days and costs | up to 12 months after randomization
  (based on Disease-Related Group codes) as a measure of health service utilization
Change in quality of life (QoL) assessed by the Cardiff Wound Impact Schedule questionnaire | from baseline to 90 days and 12 months after randomization
  Scores are transformed onto a scale of 0 - 100, a high score represents a 'good' QoL and a low score represent a 'poor' QoL
Number of patients with major amputation-free survival | up to 12 months after randomization
  death of any cause or major amputation
Number of patients with all-cause death | up to 12 months after randomization

OTHER OUTCOMES:
Infection of the index ulcer | up to 12 months after randomization
Severity of infection | up to 12 months after randomization
  defined according to Infectious Diseases Society of America (IDSA) classification
Index diabetic foot ulcer healing time | up to 12 months after randomization
  days after randomization
Change in area of the index ulcer | Compare at baseline and on 45 days, 90 days, 180 days, and 12 months after randomization
Number of patients with major adverse limb events | up to 12 months after randomization
  o Acute limb ischemia (ALI) requiring hospitalization and/ or major repeat revascularization (new bypass graft, jump/interposition graft revision, or thrombectomy / thrombolysis)
Number of patients with procedure related serious adverse events | up to 12 months after randomization
Number of patients with major bleeding | up to 12 months after randomization
  as defined by Thrombolysis in Myocardial Infarction (TIMI) Score
Number of serious adverse events | up to 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Iris Baumgartner, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (4):
- Switzerland (4):
  - Clinic for Angiology, University of Basel, Basel
  - University Clinic for Angiology, University Hospital Inselspital, Berne, Bern
  - Angiologie, Luzerner Kantonsspital, Lucerne
  - Clinic for Vascular Surgery, Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No